CLINICAL TRIAL: NCT04346615
Title: BHV3500-203: Phase 2/3: Double-Blind, Randomized, Placebo Controlled, Safety and Efficacy Trial of Zavegepant (BHV-3500) Intranasal (IN) for Hospitalized Patients With COVID-19 Requiring Supplemental Oxygen
Brief Title: Safety and Efficacy Trial of Zavegepant* Intranasal for Hospitalized Patients With COVID-19 Requiring Supplemental Oxygen
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment due to evolution of COVID-19 pandemic with reduction in patients at risk for severe disease and growing number of effective alternative therapies
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3500-203; C5301004 (Other: Alias Study Number)
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; COVID; Coronavirus; Biohaven; Intranasal; SARS-CoV-2; BHV-3500; Zavegepant
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zavegepant (Experimental): Zavegepant (BHV-3500) 10 mg intranasal (IN) dosed every 8 hours (3 times/day) (Q8h) for 14 days
  Interventions: Drug: Zavegepant (BHV-3500)
- Placebo (Placebo Comparator): Placebo Q8h for 14 days
  Subjects dosed every 8 hours; 3 times/day (Q8h)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zavegepant (BHV-3500) — 10 mg intranasal (IN) for 14 days
  Arms: Zavegepant
Drug: Placebo — Placebo Q8h for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a CGRP receptor antagonist may potentially blunt the severe inflammatory response at the alveolar level, delaying or reversing the path towards oxygen desaturation, Acute respiratory distress syndrome (ARDS), requirement for supplemental oxygenation, artificial ventilation or death in patients with COVID-19 on supplemental oxygen.

* BHV-3500, formerly "vazegepant", is now referred to as "zavegepant" (za ve' je pant). The World Health Organization (WHO) International Nonproprietary Names (INN) Expert Committee revised the name to "zavegepant" which was accepted by the United States Adopted Names (USAN ) Council for use in the U.S. and is pending formal adoption by the INN for international use.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide informed consent in accordance with requirements of the study center's institutional review board (IRB) or eithics committee prior to the initiation of any protocol-required procedures
2. Subjects must agree to provide all requested demographic information (i.e. gender, race)
3. Subjects must be able to read and understand English or Spanish
4. Subjects must be over the age of 18 years
5. Subjects must have laboratory-confirmed SARS-CoV-2 infection as determined by PCR-based commercial or public health assay
6. Subjects must have symptoms that require hospitalization with supplemental oxygen and / or non-invasive ventilation as determined by the admitting physician. The maximum nasal cannula O2 concentration should be determined by the treating clinician and the limitations of the specific equipment
7. Subjects must be willing and able to comply with study-related procedures/assessments

Exclusion Criteria:

1. Subjects in immediate need of invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
2. Subjects with an eGFR < 30 mL/min, at the Screening Visit
3. Prisoners or subjects who are involuntarily incarcerated
4. Subjects who are participating in any other investigational clinical trial while participating in this clinical trial
5. Subjects who are under the age of 18 years
6. Subjects who are pregnant (all potential female enrollees need to have a negative pregnancy test prior to IP administration)
7. Subjects with multi-organ failure
8. Subjects who have received more than 48 hours of supplemental oxygen prior to randomization
9. Subjects with prior significant pulmonary disease (e.g., severe COPD/ILD/CHF/IPF) are excluded
10. Subjects receiving investigational therapies as part of a formal clinical trial for the treatment of COVID-19. During the course of this study, investigational therapies that may become "standard of care" to treat COVID-19, but are not part of a clinical trial, are allowed
11. Subjects who are on long-acting CGRP monoclonal antibodies will be excluded including Aimovig (erenumab), Emgality (galcanezumab), Ajovy (fremanezumab), and Vyepti (eptinezumab). Additionally, the investigational oral CGRP receptor antagonist, atogepant, that is taken daily will also be excluded. Oral CGRP receptor antagonists, Nurtec ODT (rimegepant) and Ubelvy (ubrogepant) that are typically used PRN infrequently will not be excluded as long the subject was not taking them on a daily basis and does not take them during the current study
12. Subjects who are unlikely to survive for more than 48 hours from the Screening Visit
13. Subjects with any of the following abnormal laboratory values at screening: aspartate AST or ALT greater than 5x ULN or bilirubin greater than 2x ULN
14. Subjects with known active TB, history of incompletely treated TB, suspected or known extrapulmonary TB
15. Subjects with suspected or known systemic bacterial or fungal infections. However, empiric antibiotics are permitted.
16. Subjects who have participated in any clinical research study evaluating an IP or therapy within 3 months and less than 5 half-lives of IP prior to the screening visit
17. Subjects with any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject by their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Georgetown University Hospital Research Pharmacy, Washington D.C., District of Columbia
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Roper Hospital, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3500-203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 participants signed the informed consent form and were enrolled in the study, of which 3 participants failed screening and 44 participants were randomized in the study. The study was terminated early because of lack of enrollment due to the evolution of the COVID-19 pandemic, with a reduction of participants at risk for severe disease, and a growing number of effective alternative therapies.
Groups:
- Zavegepant: Participants were randomized to receive 10 milligrams (mg) of zavegepant via the intranasal route every 8 hours (± 2 hours) for approximately 14 days (42 doses) during the double-blind treatment phase. Participants had an end of treatment visit on Day 15. Participants were followed up until Day 60.
- Placebo: Participants were randomized to receive placebo via the intranasal route every 8 hours (± 2 hours) for approximately 14 days (42 doses) during the double-blind treatment phase. Participants had an end of treatment visit on Day 15. Participants were followed up until Day 60.
Period: Overall Study
Arm/Group | Zavegepant | Placebo
Started | 29 | 15
Completed | 22 | 10
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 5 | 1
Not completed — Other | 0 | 2
Not completed — Randomized not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received >=1 dose of study drug (zavegapant or placebo)
Groups:
- Zavegepant: Participants were randomized to receive 10 mg of zavegepant via the intranasal route every 8 hours (± 2 hours) for approximately 14 days (42 doses) during the double-blind treatment phase. Participants had an end of treatment visit on Day 15. Participants were followed up until Day 60.
- Total: Total of all reporting groups
Arm/Group | Zavegepant | Placebo | Total
Number analyzed (Participants) | 28 | 15 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (13.42) | 61.1 (12.41) | 55.8 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 14 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 6 | 18
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean 6 Point Ordinal Severity Rating Scale (6POSRS) Score at Day 15
Description: The 6POSRS score was used to assess severity and ranged from 1 to 6 where: 1= Death; 2= Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO), 3= Hospitalized, on non-invasive ventilation or high-flow oxygen devices; 4= Hospitalized, requiring supplemental oxygen; 5= Hospitalized, not requiring supplemental oxygen and 6= not hospitalized. A higher score indicated a better outcome.
Time Frame: Day 15
Population: Efficacy analysis set included all participants who were randomized only once and received at least one dose of study drug. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 20 | 11
Units on a scale | 5.0 (1.81) | 4.5 (1.86)

2. Secondary Outcome: Percentage of Participants With a 6-Point Severity Rating of 5 or 6, Who Were Alive and Off Supplemental Oxygen at Day 29
Description: Percentage of participants who were alive and had a 6POSRS rating of 5 (Hospitalized, not requiring supplemental oxygen) or 6 (not hospitalized) and did not use supplemental oxygen at Day 29 were reported in this outcome measure. Participants with missing 6POSRS rating at Day 29 had the last on-study 6POSRS rating before Day 29 used. Participants with >= 1 procedure day of supplemental oxygen use before Day 29 for an ongoing procedure were considered failures, i.e., not alive or not off of oxygen at Day 29. 95% confidence interval (CI) was based on exact Clopper and Pearson method.
Time Frame: Day 29
Population: Efficacy analysis set included all participants who were randomized only once and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Percentage of participants | 67.9 [47.7 to 84.1] | 60.0 [32.3 to 83.7]

3. Secondary Outcome: Percentage of Participants With a 6-Point Severity Rating of 2 or 3 or Required Initiation of Invasive Mechanical Ventilation, Non-Invasive Ventilation, or a High-Flow Nasal Cannula Through Day 29
Description: Percentage of participants who had a 6POSRS rating of 2 (Hospitalized, on invasive mechanical ventilation or ECMO) or 3 (Hospitalized, on non-invasive ventilation or high-flow oxygen devices) or >= 1 procedure day of ventilation or high-flow nasal cannula use on study through Day 29 were reported in this outcome measure. Participants with missing 6POSRS rating at Day 29 had all available on-study 6POSRS ratings before Day 29 used. 95% CI was based on exact Clopper and Pearson method.
Time Frame: Up to Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Percentage of participants | 46.4 [27.5 to 66.1] | 60.0 [32.3 to 83.7]

4. Secondary Outcome: Percentage of Participants Admitted Into an Intensive Care Unit (ICU) Through Day 29
Description: Percentage of participants admitted into an ICU on any day through Day 29 were reported in this outcome measure. 95% CI was based on exact Clopper and Pearson method
Time Frame: Up to Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Percentage of participants | 25.0 [10.7 to 44.9] | 20.0 [4.3 to 48.1]

5. Secondary Outcome: Number of Participants With On-Treatment Deaths, Serious Adverse Events (SAEs) and Severe Adverse Events (AEs)
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. An SAE was any untoward medical occurrence that at any dose: resulted in death; was life-threatening; required prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect; other important medical events. Severe AEs were AEs that interrupted usual activities of daily living, significantly affected clinical status, or required intensive therapeutic intervention. On-treatment was defined as the time on study drug.
Time Frame: From first dose of study treatment on Day 1 until Day 15
Population: Safety analysis set included all participants who received >=1 dose of study drug (zavegapant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Participants
  Death | 1 | 1
  SAEs | 6 | 2
  Severe AEs | 7 | 3

6. Secondary Outcome: Number of Participants With Grade 3 or 4 On-Treatment Laboratory Test Abnormalities
Description: The following laboratory parameters were assessed: eosinophils, hemoglobin, leukocytes, lymphocytes (high and low), neutrophils, platelets, alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, bilirubin, calcium (high and low), creatine kinase, creatinine, glomerular filtration rate (GFR) estimated Modification of Diet in Renal Disease (MDRD), glucose (high and low), lactate dehydrogenase, potassium (high and low), sodium (high and low), urate, glucose (urine) and protein (urine). Laboratory abnormalities were graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5 for all parameters except glucose and uric acid. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 was used for grading glucose and uric acid. Grade 3=severe and grade 4=potentially life threatening. Number of participants with grade 3 or 4 laboratory abnormalities is reported.
Time Frame: From first dose of study treatment on Day 1 until Day 15
Population: Safety analysis set included all participants who received >=1 dose of study drug (zavegapant or placebo). Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Participants
  Eosinophils | 0 | 0
  Hemoglobin | 2 | 0
  Leukocytes | 0 | 0
  Lymphocytes, high | 0 | 0
  Lymphocytes, low | 3 | 3
  Neutrophils | 0 | 1
  Platelets | 0 | 0
  Alanine Aminotransferase: number analyzed (Participants) | 25 | 14
  Alanine Aminotransferase | 0 | 0
  Albumin: number analyzed (Participants) | 27 | 14
  Albumin | 1 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 25 | 14
  Alkaline Phosphatase | 0 | 0
  Aspartate Aminotransferase: number analyzed (Participants) | 25 | 14
  Aspartate Aminotransferase | 0 | 0
  Bicarbonate: number analyzed (Participants) | 28 | 14
  Bicarbonate | 0 | 0
  Bilirubin: number analyzed (Participants) | 25 | 14
  Bilirubin | 0 | 0
  Calcium, high: number analyzed (Participants) | 27 | 14
  Calcium, high | 0 | 0
  Calcium, low: number analyzed (Participants) | 27 | 14
  Calcium, low | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 22 | 14
  Creatine Kinase | 1 | 0
  Creatinine: number analyzed (Participants) | 28 | 14
  Creatinine | 1 | 1
  Glomerular Filtration Rate, Estimated MDRD: number analyzed (Participants) | 28 | 14
  Glomerular Filtration Rate, Estimated MDRD | 1 | 1
  Glucose, high: number analyzed (Participants) | 28 | 14
  Glucose, high | 5 | 2
  Glucose, low: number analyzed (Participants) | 28 | 14
  Glucose, low | 0 | 0
  Lactate Dehydrogenase: number analyzed (Participants) | 25 | 14
  Lactate Dehydrogenase | 0 | 0
  Potassium, high: number analyzed (Participants) | 28 | 14
  Potassium, high | 0 | 0
  Potassium, low: number analyzed (Participants) | 28 | 14
  Potassium, low | 0 | 0
  Sodium, high: number analyzed (Participants) | 28 | 14
  Sodium, high | 0 | 0
  Sodium, low: number analyzed (Participants) | 28 | 14
  Sodium, low | 1 | 0
  Urate: number analyzed (Participants) | 24 | 12
  Urate | 0 | 0
  Glucose, Urine: number analyzed (Participants) | 7 | 3
  Glucose, Urine | 0 | 0
  Protein, Urine: number analyzed (Participants) | 7 | 3
  Protein, Urine | 0 | 0

7. Secondary Outcome: Number of Participants With Severe or Life-Threatening Bacterial, Invasive Fungal, or Opportunistic Infections Through Day 29
Description: Number of participants with any severe or life-threatening bacterial, invasive fungal, or opportunistic infections through Day 29 is reported in this outcome measure. Severe= interrupted usual activities of daily living, significantly affected clinical status, or required intensive therapeutic intervention. Life threatening=Participant was at immediate risk of death from the event as it occurred; i.e., it did not include a reaction that if it had occurred in a more serious form might have caused death.
Time Frame: Up to Day 29
Population: Safety analysis set included all participants who received >=1 dose of study drug (zavegapant or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants were randomized to receive placebo via the intranasal route every 8 hours (± 2 hours) for approximately 14 days (42 doses) during the double-blind treatment phase. Participants had an end of treatment visit on Day 15. Participants were followed up until Day 60. Participants were followed up until Day 60.
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Participants | 5 | 1

8. Secondary Outcome: Number of Participants With Intranasal Administration Reactions Through Day 29
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational product and that did not necessarily have a causal relationship with this treatment. Number of participants with any adverse events associated with intranasal administration were reported in this outcome measure.
Time Frame: Up to Day 29
Population: Safety analysis set included all participants who received >=1 dose of study drug (zavegapant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 15
Participants | 16 | 3

9. Secondary Outcome: Percentage of Participants With >= 50% Reduction in Estimated Glomerular Filtration Rate (eGFR) From Baseline
Description: Percentage of participants with >=50% reduction in eGFR from Baseline during on-treatment phase were reported in this outcome measure.
Time Frame: From Baseline (Day 1) up to Day 15
Population: Safety analysis set included all participants who received >=1 dose of study drug (zavegapant or placebo). Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 28 | 14
Percentage of participants | 7.1 | 14.3

ADVERSE EVENTS:
Time Frame: On treatment: From start of study drug on Day 1 up to Day 15 and Follow up: From Day 16 to Day 60
Description: Same event may appear as both an SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Groups:
- Zavegepant (On-treatment): Participants received 10 mg of zavegepant via the intranasal route every 8 hours (± 2 hours) for approximately 14 days (42 doses) during the double-blind treatment phase.
- Placebo (On-treatment): Participants received placebo via the intranasal route every 8 hours (± 2 hours) for approximately 14 days (42 doses) during the double-blind treatment phase.
- Zavegepant (Follow-up): Participants who received zavegepant during the double-blind treatment phase were followed up from Day 16 to Day 60.
- Placebo (Follow-up): Participants who received placebo during the double-blind treatment phase were Followed up from Day 16 to Day 60.
Arm/Group | Zavegepant (On-treatment) | Placebo (On-treatment) | Zavegepant (Follow-up) | Placebo (Follow-up)
All-Cause Mortality (participants affected / at risk) | 1/28 | 1/15 | 4/27 | 0/13
Serious Adverse Events (participants affected / at risk) | 6/28 | 2/15 | 2/27 | 1/13
Other Adverse Events (participants affected / at risk) | 22/28 | 13/15 | 4/27 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Zavegepant (On-treatment) (N=28) | Placebo (On-treatment) (N=15) | Zavegepant (Follow-up) (N=27) | Placebo (Follow-up) (N=13)
Endotracheal intubation (Surgical and medical procedures) | 3 | 2 | 0 | 0
Intensive care (Surgical and medical procedures) | 3 | 0 | 0 | 0
Gastrostomy tube removal (Surgical and medical procedures) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0/13 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant (On-treatment) (N=28) | Placebo (On-treatment) (N=15) | Zavegepant (Follow-up) (N=27) | Placebo (Follow-up) (N=13)
Dysgeusia (Nervous system disorders) | 16 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 8 | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Intensive care (Surgical and medical procedures) | 4 | 3 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 2 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 1 | 2 | 0 | 0
Transaminases increased (Investigations) | 1 | 2 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Scleral oedema (Eye disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04346615/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04346615/SAP_001.pdf